CLINICAL TRIAL: NCT01907464
Title: Physiopathology of Bone Loss in Young Patient With Anorexia Nervosa
Brief Title: Bone Loss in Patients With Anorexia Nervosa
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: UF 8751
Record Dates: First submitted 2013-07-17; First posted 2013-07-25 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Patients With Anorexia Nervosa
Keywords: Anorexia nervosa; Bone mineral density; Teenagers or young women; Bone remodelling markers
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients with anorexia nervosa (Experimental): This arm is the experimental arm composed of patients
  Interventions: Other: clinical parameters description; Other: para clinical parameters description; Other: hormonal parameters dosing; Other: bone modeling markers dosing
- controls subjects (Active Comparator): This arm is composed of healthy volunteers
  Interventions: Other: clinical parameters description; Other: para clinical parameters description; Other: hormonal parameters dosing; Other: bone modeling markers dosing

INTERVENTIONS:
Other: clinical parameters description — description of weight, height, Bone Mass Index, dietary questionnary, amenorrhea time, pathology time for the two arms
Other: para clinical parameters description — description of DMO, mass, basal metabolism, IGF-1/IGFBP-3 for the two arms
Other: hormonal parameters dosing — dosing of leptine, leptine receptor, adiponectine, ghreline for the two arms
Other: bone modeling markers dosing — dosing of osteocalcine, bone alkalin phosphatase, C-telopeptide of type-I collagene, osteoprotegerine/ RANKL for the two arms

SUMMARY:
Nutritional deprivation of adolescent girls with anorexia nervosa (AN) reduces the bone mass acquisition. A better understanding of this process would improve the medical treatment of bone alteration and its long-term consequences.

160 patients (age < 38 yr) with AN and 160 age-matched controls (CON) will be enrolled in this study. The areal bone mineral density (aBMD) will be determined using dual-X-ray absorptiometry. Calciotropic hormones, bone turnover markers will be concomitantly evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Health Insurance regimen or benefit from an health insurance regimen
* Aged from 14 to 38 years old
* Women
* No pregnant

Specific inclusion criteria for patient:

Patient suffering from anorexia nervosa defined by criteria of Diagnostic and Statistical Manual of Mental Disorders (DSM-IV)

Specific inclusion criteria for controls:

* Normal menstrual cycles,
* No lifetime history of eating disorders,
* BMI between 18 and 25 kg/m²

Exclusion Criteria:

* use of treatments may be modify bone mass (bisphosphonates,…)
* Disease or treatment may be induce osteoporosis
* In exclusion period in relation with another study
* Law protected subject

Ages: 14 Years to 38 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 320 (Estimated)
Dates: Start 2011-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Dual-X-ray absorptiometry (DEXA) | at Day 0 (time of the inclusion visit)
  The primary outcome is to model the bone mass acquisition in young women with anorexia nervosa.

SECONDARY OUTCOMES:
Biological parameters identification | At day 0 (time of the inclusion visit)
  One of the secondary outcome is to identify biological factors associated with bone demineralisation.
clinical parameters identification | At Day 0 (at time of the the inclusion visit)
  One of the secondary outcome is to identify the clinical factors associated with bone demineralisation.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick PL LEFEBVRE, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- CHU de Montpellier - Département d'Endocrinologie Diabète, Montpellier, France